CLINICAL TRIAL: NCT07156279
Title: The Effect of Emotional Freedom Technique (EFT) Applied to Pregnant Women Before Cesarean Delivery on Surgical Fear and Intra-operative Vital Signs
Brief Title: Effect of Emotional Freedom Technique on Surgical Fear and Vital Signs in Women Undergoing Cesarean Section
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Derya Bingöl, LECTURER, Bingol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BINGOL UNİVERSİTY
Record Dates: First submitted 2025-04-07; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section; Preoperative Anxiety
Keywords: Emotional Freedom Techniques (EFT); Intraoperative Hemodynamics; Apgar Score; Surgical Fear; Cesarean Delivery

STUDY DESIGN:
Intervention Model Description: Emotional Freedom Technique-EFT EFT basically involves clicking and touching acupuncture points, needles are not used, there is no invasive intervention, there are affirmation suggestions, it is an easy, painless, simple but effective method that can be done in minutes. Many studies have shown that in addition to the insertion of acupuncture needles, acupuncture stimulation can also be provided by vacuum suction, touching, ultrasound and acupressure, and randomized controlled studies have shown that somatic stimulation (acupressure) has the same effect as needles. (Craig, 2004) It is performed by applying kinetic energy to certain meridians on the head and chest with the fingertips. The points where the tapping is done are the end points of the meridians in the body. They are located symmetrically on both sides of the body. Since these points are close to the skin surface, they are points that are more easily reached than the deeper buried parts of the meridians.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT (Emotional Freedom Technique) (Experimental): Participants in the experimental group will receive Emotional Freedom Technique (EFT) sessions lasting 15-20 minutes. EFT is a behavioral intervention in which individuals tap with their fingertips on specific acupressure points on the head and chest while focusing on a target issue. The technique is non-invasive, painless, and simple to apply. Sessions also include the use of positive affirmations during tapping.
  Interventions: Behavioral: EFT(Emotional Freedom Technique)
- Control Group (No Intervention): No intervention will be applied to participants in the control group. They will complete study questionnaires and receive routine information only.

INTERVENTIONS:
Behavioral: EFT(Emotional Freedom Technique) — EFT is a behavioral intervention in which participants tap with their fingertips on specific acupressure points while focusing on a target issue. The technique is non-invasive, painless, and simple to apply. Sessions also include the use of positive affirmations during tapping.
  Other Names: Emotional freedom technique; EFT
  Arms: EFT (Emotional Freedom Technique)

SUMMARY:
Surgical interventions are unusual interventions that can cause anxiety and fear in individuals. It is known that anxiety and fear experienced during this period affect the intraoperative and postoperative process. Emotional Freedom Technique (EFT) is a type of energy psychotherapy that has no side effects and its effect on fear has been demonstrated in many studies. This study will be conducted to determine the effect of Emotional Freedom Technique (EFT) applied in the preoperative period in pregnant women planned to have a cesarean section on surgical fear, intraoperative hemodynamics and newborn Apgar score.

Research questions:

1. Does EFT Technique reduce surgical fear level?
2. Does EFT Technique affect intraoperative hemodynamics?
3. Is EFT Technique effective on newborn Apgar score?
4. Is there a relationship between surgical fear and intraoperative hemodynamics and newborn Apgar score? The research will be conducted in two stages in the Gynecology and Obstetrics Department of Bingöl State Hospital and the operating room unit of the same hospital. The universe of the study will consist of women who are scheduled for elective cesarean delivery and who do not have a risky pregnancy and who are admitted to Bingöl State Hospital. Considering the possibility of data loss due to various reasons during the study process, it is planned to be completed on a total of 60 women, 30 in the experimental group and 30 in the control group.

DETAILED DESCRIPTION:
Surgical interventions are often performed to secure people's lives. Although these applications are routine procedures for health professionals, exposure to a medical or surgical intervention in the operating room environment is a stress factor as it is unusual for most patients . Studies show that patients waiting for surgical intervention experience intense fear, anxiety, and anxiety in the preoperative period and that this is a situation that is often ignored .

Studies indicate that younger patients have higher anxiety levels than older patients and female patients have higher anxiety levels than male patients. Again, the results of some studies examining the factors causing anxiety and fear suggest that obstetric surgeries may cause more anxiety in individuals than some other surgeries .

Cesarean section (C/S) delivery represents one of the most common surgical interventions, which has increased significantly in many parts of the world in recent years .Cesarean section (C/S) rates are increasing worldwide, making C/S the most common intraperitoneal surgical intervention . According to Turkish population and health survey 2018 data, the cesarean section rate in our country is 52%, which is unfortunately much higher than the cesarean section rate recommended by WHO (World Health Organization). Again, one in three women in the United States gives birth by cesarean section, making C/S one of the most common surgical procedures in the country. The fact that caesarean section rates have increased so much in all countries of the world, developed and developing alike, should support efforts to reduce this method of delivery and promote normal delivery methods, but should also aim to minimize the side effects of this surgical procedure and the accompanying anesthesia and focus equally on postoperative maternal and fetal health outcomes.

The anxiety and fear experienced by pregnant women before these surgical interventions, the frequency of which has increased considerably in all countries of the world, are often ignored for various reasons, as in other surgeries. However, in addition to the fear and anxiety caused by surgical intervention in pregnant women before this intervention, the problems that may occur in the baby to be born are an additional cause of fear and anxiety. The results of the studies suggest that preoperative emotional states and fears of the patients should be determined and appropriate interventions should be made, since the preoperative emotional states and fears of the patients will affect compliance with the surgical process.

In C/S operations, spinal anesthesia technique is preferred in the first place due to its ease of application.Although spinal anesthesia provides significant benefits compared to general anesthesia, it often leads to hypotension with an incidence of up to 60% to 70% due to sympathetic nervous system blockade . Hypotension after spinal anesthesia is a common complication that can have adverse effects on the well-being of both the laboring woman and the fetus . Prolonged hypotension leads to cardiovascular problems and additional organ damage. At the same time, decreased placental blood flow in utero leads to fetal hypoxia, acidosis, and thus affected fetal health and lower Apgar scores. Since intraoperative hypotension is associated with increased patient morbidity, it is very important to maintain hemodynamics in cesarean section operations, especially in the perinatal period before fetal delivery.

Maternal hypotension after spinal anesthesia is mainly due to blockade of sympathetic efferent neurons. Studies have shown that patients with higher basal sympathetic activation have more pronounced hypotension after spinal anesthesia . Anxiety and fear, which are often experienced in patients in the preoperative period, also cause general sympathetic activation. These findings provide us with a rational basis for the hypothesis that hypotension may become more pronounced after induction of spinal anesthesia in pregnant women with high anxiety levels in the preoperative period.

Benzodiazepines are used as classical therapeutic agents in the management of surgical fear and anxiety, which are intensely experienced in the preoperative period and have been shown to have a serious effect on postoperative patient outcomes by many studies . Due to the post-op complications of benzodiazepines (delirium, mortality, morbidity, etc.), the routine use of these drugs and the reduction of their use have been frequently discussed in recent years. The European Society of Anesthesiology and Intensive Care also recommends avoiding routine premedication with benzodiazepines . The use of complementary methods such as supportive talks, acupuncture, aroma therapy and relaxation methods, music recital, etc. instead of pharmacological treatments in the management of preoperative surgical fear and anxiety has become a focus .

Energy is in constant flow in the human body and all humans have an energy body. Blockages/problems that occur in our body prevent the flow of energy. As a result, the balance between mind/body/energy is disrupted.. EFT is an easily applicable type of energy psychotherapy. The basic principle of evidence-based EFT applications, which are highly effective and successful in clinical problems, is that individuals' limiting or disturbing emotions and thoughts disrupt the energy flow in the body and create blockages in energy points .

Emotional Freedom Technique (EFT) is a type of energy psychotherapy with no side effects and its effect on fear has been demonstrated in many studies. This study will be conducted to determine the effect of EFT on surgical fear, intraoperative hemodynamics and neonatal apgar score in pregnant women who are scheduled for cesarean delivery.

The place and characteristics of the research The research will be conducted in two stages in Bingöl State Hospital Obstetrics and Gynecology service and the operating room unit of the same hospital. At Bingöl State Hospital, where 8 gynecologists are currently working, an average of 120 women are delivered by cesarean section on a monthly basis and 4 women on a daily basis.

The population of the study will consist of women without risky pregnancies who applied to Bingöl State Hospital and planned elective delivery by cesarean section. Which participants will be included in the intervention and control groups was determined by randomization on www.random.org. . Considering the possibility of data loss due to various reasons during the research process, it was planned to be completed on a total of 60 women, 30 experimental and 30 control groups.

Data Collection Tools Descriptive Characteristics Form It is a form prepared by the researcher by reviewing the literature and includes the sociodemographic characteristics of the participants (age, height, weight, occupation, family type, education level, income level, etc.).

Subjective Units of Experience (SUE) Scale:

Using the SUE chart or SUE scale, a subjective scoring of the current emotion or experience is made. With the scoring on the SUE scale, it provides us with concrete data about the effectiveness of the process, both the score given to the current emotion before EFT and the scoring after EFT. On the scale from "-10" to "+10", the person rates the emotion that disturbs them such as fear, anxiety, distress Pre-Op Vital Signs Follow-up Form It is a form prepared by the researcher that allows the vital signs (blood pressure, pulse, respiration) of the patients in the preoperative period to be recorded before and after the intervention.

Surgical Fear Scale:

Consisting of 8 items, the scale is an 11-point Likert scale scored between 0-10. Each item in the scale is scored as 0 "not at all afraid" and 10 "very afraid".

The scale has two sub-dimensions, each consisting of four items. These sub-dimensions show the fear of short-term and long-term consequences of the surgery. Items 1-4 measure fear of short-term consequences of surgery, while items 5-8 measure fear of long-term consequences of surgery. The total score of the scale is minimum 0 and maximum 80 points. The higher the score, the higher the level of surgical fear.

Hemodynamic Parameters Record Form It is a form prepared by the researchers by reviewing the literature to record hemodynamic findings (HR, SPO2, BP, fluid balance, amount of bleeding, etc.) and neonatal apgar scores in the intraoperative period.

Data Collection The data will be collected between February 2025 and June 2025 on weekdays when cesarean section operations are mostly performed in the Gynecology Department of Bingöl State Hospital. Data collection will be in two stages. The data in the first stage will be collected face-to-face by one of the researchers in the patient room after the patients are hospitalized in the ward on the day they will be operated in the pre-op period. Patients in the control group will be administered the Descriptive Characteristics Form, SUE scale, Surgical Fear Scale, without any intervention other than the clinical protocol, and their pre-op vital signs will be recorded. Surgical Fear Scale will be applied again after 30 minutes without any intervention other than routine cesarean section preop preparation practices to pregnant women whose vital signs are taken. For the patients in the experimental group who will be applied emotional liberation technique; just before the emotional liberation technique session; Descriptive Characteristics Form, Surgical Fear Scale and SUE scale will be applied and routine pre-op preparations will be expected to be completed after the vital signs are measured. Then, the Emotional Freedom Technique (EFT) will be applied by the researcher who has an Emotional Freedom Technique Practitioner certificate for a session lasting approximately 20 minutes. After the session, the SUE scale and then the Surgical Fear Scale will be administered again without a break. In Phase 2 of the study, the other researcher will record the vital signs, other hemodynamic parameters and neonatal apgar score of the patients who are operated for cesarean section by using the Hemodynamic Parameters Recording Form during the operation without knowing which patient is in the experimental group and which patient is in the control group.

Nursing Initiative (Phase 1) (EFT) EFT basically involves clicking and tapping on acupuncture points, no needles, no invasive intervention, affirmation suggestion sentences, and is an easy, painless, simple but effective method that can be done in minutes.

While applying pressure with the fingertips, the person should concentrate on whatever is bothering them. Another thing to do at the same time is to make positive suggestions to oneself out loud.

Tapping Points Emotional frredom technique will be practiced by a trained researcher in the quietest and calmest environment possible, in a position where the patient is comfortable. Initially, the patient will be asked to focus on his/her fear, to recognize the discomfort he/she feels and to express his/her problem out loud (e.g. I am worried about having surgery, I am very afraid of having surgery). The patient will then be asked to evaluate the discomfort she feels due to fear with the SUE Scale, which is the first stage of the Emotional Freedom Technique, and to give a score. The pregnant woman will be asked to say the set-up sentence (I accept myself completely and as I am, even though I am anxious, nervous and afraid) and repeat the sentence three times and then the acupuncture points will be tapped (each acupuncture point should be tapped 7-8 times with the fingertips). At this stage, the patient will be asked to repeat the sentence (this fear, this worry, this anxiety, this concern) briefly (this is also called a reminder sentence). The tapping will start at the vertex on the top of the pregnant woman's head. Then, the strokes will be applied to the starting points of both eyebrows, which the researchers call the eyebrow points. After the corners of the eyes, under the eyes, under the nose, under the lips, the CB point (2.5-3 cm below the junction of the breastbone and collarbone and 2.5-3 cm to the right or left) will be followed by strokes on the fingers of the right and left hand - thumb, index finger, middle finger, little fingers, respectively. Immediately after the last finger of each hand is tapped, the karate point, which is the fleshy outer side of the hand following the little finger, is tapped so that the pregnant woman can hear the sentences. While tapping each point from the top of the head to the karate point, the pregnant woman will be asked to repeat the set-up sentence or reminder sentences. Between the two points, the pregnant woman will be asked to take a deep breath first. After one round is over, the heart will be moved to the healing position and she will be asked to score her fear and anxiety again according to the SUE ScaleINTRA-OP DATA COLLECTION (Phase 2) In the second phase of the study, pregnant women who were admitted to the operating room for CS operation were taken to the premedication room by the other investigator without knowing which of the experimental and control groups they were in. Pregnant women whose general evaluation was not suitable for spinal anesthesia were excluded from the study, and only pregnant women who were decided to undergo spinal anesthesia were recorded using a follow-up form. Spinal anesthesia will be administered with 2.2-2.8 mL (11-14 mg) 0.5% hyperbaric bupivacaine according to the patient's height and weight. Immediately after routine intrathecal injection of local anesthetic, hemodynamic data such as cardiac heart rate (HR), oxygen saturation (SPO2), systolic arterial pressure (SBP), diastolic arterial pressure (DBP), mean arterial pressure (MAP) values, amount of inotropic and sedative agents to be used intraoperatively, baseline, in the sitting position before spinal block, immediately after subarachnoid injection (0. min), at 1st, 3rd, 6th, 9th, 12th, 15th min, immediately after delivery, at 10 min intervals after delivery and at recovery exit will be recorded on the Hemodynamic Parameters Record Form.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteer to participate in the study,
* Those who can understand and speak Turkish,
* Those who are ASA II in the American Anesthesiologists Association risk classification,
* Pregnant women who will undergo elective CS,
* Women without a risky pregnancy (gestational diabetes mellitus, preeclampsia, eclampsia, HT patients, CHD, etc., multiple pregnancy, pregnancy with in vitro treatment),
* Pregnant women between the ages of 20-40,
* Pregnant women without any psychiatric comorbidities,
* Pregnant women with a Fear score below 0 according to the SUE Scale. (Pregnant women who state that they are afraid of surgical procedures)

Exclusion Criteria:

* Those with serious heart, lung, liver disease, kidney failure, bleeding diathesis, fever, infection, allergy to the drugs to be used,
* Patients with hypothermia and acid-base disorders and electrolyte disorders,
* Those taking antibiotics, anticonvulsants, antiarrhythmics, cholinesterase inhibitors,
* Pregnant women who decide to undergo general anesthesia for various reasons,
* Pregnant women at risk,

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since pregnant women scheduled for cesarean delivery will be included in the study, individuals whose biological sex is female will be included.
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Surgical Fear Score (Surgical Fear Scale, total) | From baseline preoperative assessment on the day of surgery (after hospital admission and before EFT application) to thirty minutes after the EFT session, within the same preoperative day before transfer to the operating room.
  Change in the total score of the 8-item Surgical Fear Scale (range 0-80; each item scored 0-10). Scores will be assessed before and immediately after the EFT session in the intervention group, and at equivalent time points in the control group. Reporting will be done as the change score between the two time points and/or as a percentage change.

SECONDARY OUTCOMES:
Intraoperative Heart Rate (HR) | From intraoperative baseline before spinal anesthesia until recovery room exit on the same operative day.
  Average heart rate during the intraoperative period and its course over time (at predefined time points).
Intraoperative Blood Pressure (systolic, diastolic, mean arterial pressure) | From intraoperative baseline before spinal anesthesia until recovery room exit on the same operative day.
  Intraoperative measurements of systolic, diastolic, and mean arterial pressure values at predefined time points.
Intraoperative Oxygen Saturation (SpO₂) | From intraoperative baseline (before spinal anesthesia and zero minutes after intrathecal injection) until recovery room exit on the same operative day.
  Intraoperative oxygen saturation measurements; minimum SpO₂ and mean SpO₂.
Incidence of Intraoperative Hypotension | From intraoperative baseline (before spinal anesthesia and zero minutes after intrathecal injection) until recovery room exit on the same operative day.
  Incidence of intraoperative hypotension. Recommended definition: SBP < 90 mmHg or ≥20% decrease from baseline; at least one occurrence is considered present.
Use of Vasopressors During Surgery | From intraoperative baseline (before spinal anesthesia and zero minutes after intrathecal injection) until recovery room exit on the same operative day.
  Vasopressor use during surgery (yes/no) and number of applications (bolus number) recorded in the Anesthesia record form
Estimated Blood Loss (EBL) | From intraoperative baseline (before spinal anesthesia and zero minutes after intrathecal injection) until recovery room exit on the same operative day.
  Estimated amount of intraoperative bleeding.Surgical/anesthesia records (gas buffer count method)
Apgar Score at 1 and 5 minutes | In the 1st and 5th minutes after birth
  Apgar scores of the newborn at 1 and 5 minutes.
Change in Subjective Units of Experience (SUE) Score | Between two preoperative measurements (same day, before surgery).
  Change in Subjective Units of Experience (SUE) Scale score. This is a subjective self-rating scale that ranges from -10 to +10, where -10 represents the most negative distress and +10 represents the most positive emotional state. Higher scores indicate a better emotional state (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl Üniversitesi, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of individual participant data is being considered